CLINICAL TRIAL: NCT00950053
Title: Chronic Insertional Achilles Tendonitis Treated With or Without Flexor Hallucis Longus Tendon Transfer: A Prospective, Randomized, Controlled Trial
Brief Title: Chronic Insertional Achilles Tendonitis Treated With or Without Flexor Hallucis Longus Tendon Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120808A
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Insertional Achilles Tendonitis
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Achilles decompression & debridement (Active Comparator)
  Interventions: Procedure: Achilles decompression & debridement
- Achilles decompression,debride&FHLtransf (Active Comparator): Achilles tendon decompression and debridement augmented with FHL transfer. The preferred skin incision will be followed by central-splitting Achilles debridement, resection of a Haglund's lesion if present and pathologic, followed by FHL harvest for patients in group 2. The fixation technique in group 2 will utilize an interference screw for the FHL. For all patients, the Achilles will be reattached with lateral and medial suture anchors (just distal to interference screw in FHL patients).
  Interventions: Procedure: Achilles decompression and debridement with FHL transfer

INTERVENTIONS:
Procedure: Achilles decompression & debridement — Surgical intervention
  Arms: Achilles decompression & debridement
Procedure: Achilles decompression and debridement with FHL transfer — surgical intervention
  Arms: Achilles decompression,debride&FHLtransf

SUMMARY:
The purpose of this study is to determine whether Achilles tendon debridement and decompression augmented with flexor hallucis longus (FHL) tendon transfer results in improved clinical and functional outcome as measured by ankle plantar flexion strength and American Orthopedic Foot and Ankle Society (AOFAS) score compared to debridement and decompression alone in patients over 50 years of age with chronic insertional Achilles tendinosis.

H0: There will be no difference in ankle plantar flexion strength measured using a handheld dynamometer between patients randomized to achilles tendon decompression and debridement alone (Group 1) and patients randomized to achilles tendon decompression and debridement augmented with FHL transfer (Group 2).

HA: Patients randomized to achilles tendon decompression and debridement alone (Group 1) will have less ankle plantar flexion strength compared to patients randomized to achilles tendon decompression and debridement augmented with FHL transfer (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years of age or older
* Patients diagnosed with chronic insertional Achilles tendonitis
* Failed greater than 3 months of conservative treatment (activity and shoe modification, heel lifts, non-steroidal anti-inflammatory medications, stretching exercises, and formal physical therapy)

Exclusion Criteria:

* Patients less than 50 years of age upon presentation
* Females of child-bearing potential
* Patients who have a history of ipsilateral Achilles tendon rupture
* History of infection in the same lower extremity
* Patients unable to undergo MRI scan

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
ankle plantar flexion strength measured using a handheld dynamometer | pre-operatively, 3 months, 6 months, and 1 year

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society(AOFAS) Ankle-Hindfoot score | pre-operatively, 3 months, 6 months, and 1 year
Visual analog pain scale (VAS) | pre-operatively, 3 months, 6 months, and 1 year
Hallux plantarflexion strength using the dynamometer | pre-operatively, 3 months, 6 months, and 1 year
Patient Satisfaction | 1 year
Surgical complications | Date of Surgery
Postoperative complications | 3 months, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Cohen, MD, Principal Investigator — OrthoCarolina, P.A.
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States